CLINICAL TRIAL: NCT06100302
Title: The First Afﬁliated Hospital of Xi'an Jiaotong University
Brief Title: Study on the Mechanism of Immune Inflammation in Cognitive Impairment of Depression
Acronym: depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-249
Record Dates: First submitted 2023-09-17; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Depression
Keywords: depression; Immune metabolism; Cognitive function
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MD group: Patients with depression who met the inclusion criteria
  Interventions: Other: no-intervention
- HC group: Healthy subjects meeting enrollment criteria
  Interventions: Other: no-intervention

INTERVENTIONS:
Other: no-intervention — no-intervention

SUMMARY:
The patients with depression were observed and followed up to evaluate the changes of symptoms and cognitive function in patients with depression at different time points before and after drug treatment. At the same time, immunometabolism indicators in serum, urine and stool were detected to screen out immunoinflammatory markers related to cognitive function and treatment response in patients with depression, hoping to provide a new strategy for optimal treatment of depression.

DETAILED DESCRIPTION:
1. Participants were included according to the inclusion and exclusion criteria, and demographic data of depressed patients and healthy controls were recorded, including age, sex, ethnicity, occupation, etc. Subjects in the depression group were treated with antidepressants (as recommended by the guidelines) and were followed up baseline, 2 weeks, 8 weeks, 12 weeks, and 24 weeks after treatment, respectively. At each follow-up point, symptoms were assessed using Hamilton Depression Scale (HAMD), Hamilton Anxiety Scale (HAMA), Depression Screening Scale (PHQ-9) and Generalized Anxiety Scale (GAD-7), and cognitive function was assessed using Thinc-it at three follow-up points: baseline, 12 weeks after treatment, and 24 weeks after treatment. General data were compared between patients with depression and healthy controls at baseline.
2. The depression group was followed up. Serum and fecal of patients with depression were collected at 5 follow-up points at baseline, 2 weeks, 8 weeks, 12weeks and 24 weeks after treatment, and serum metabolic indexes and fecal metagenome were detected.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old, male or female;
* Meet the diagnostic criteria for depression in the International Classification of Diseases-10 (ICD-10), and the Hamilton Depression Scale (HAMD) score ≥18 points;
* Junior high school education and above, can cooperate with the completion of relevant scales and sample collection;
* did not receive antidepressant therapy at admission or took medication for less than 14 days; And the duration of drug withdrawal ≥3 months;
* No history of infection and taking hormones, antibiotics or anti-inflammatory drugs in the past 1 month;
* History of physical diseases such as centerless, liver, kidney and gastrointestinal tract, active infection, active or chronic inflammation, autoimmune diseases, etc.

Exclusion Criteria:

* Pregnant and lactating women;
* Clinically significant or unstable medical conditions, including congestive heart failure, liver and kidney failure, cancer, immune and metabolic endocrine diseases;
* Patients with acute or chronic infection, taking anti-inflammatory drugs, cortisol hormones, and receiving antibiotics for 3 consecutive days in the past 1 month;
* Patients with neuropsychiatric diseases other than depression.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Meet the diagnostic criteria for depression in the International Classification of Diseases-10 (ICD-10), and the Hamilton Depression Scale (HAMD) score ≥18 points
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Scores of Hamilton Depression Scale | baseline、2weeks、8weeks、12weeks、24weeks
  Using to assess depressive symptoms. With higher scores associated with more severe depression symptoms. Total scores <7 is normal; Mild depression with total scores of 7～17; Moderate depression with total scores of 18～24; Total scores >24 for severe depression.
Scores of Hamilton Anxiety Scale | baseline、2weeks、8weeks、12weeks、24weeks
  Using to assess anxiety symptoms. With higher scores associated with more severe anxiety symptoms. Total scores< 7 indicates no anxiety; Total scores≥7 indicates possible anxiety; Total scores≥14 indicates anxiety; Total scores≥21 indicates obvious anxiety; Total scores≥29 points indicates serious anxiety.
Patient Health Questionnaire-9 | baseline、2weeks、8weeks、12weeks、24weeks
  Using to assess depression symptoms, scores range from 0～27, With higher scores associated with more severe depression symptoms. Total scores 0～4 indicates no depression; Total scores 5～9 indicates mild depression; Total scores 10～14 indicates moderate depression; Total scores 15～19 indicate moderate to severe depression; Total scores 20～27 indicates major depression.
Generalized self-rating anxiety Scale | baseline、2weeks、8weeks、12weeks、24weeks
  Using to assess anxiety symptoms, scores range from 0～21. With higher scores associated with more severe anxiety symptoms. Total scores 5～9 indicates mild anxiety; Total scores 10～14 scores indicate moderate anxiety; Total scores 15～21 scores indicate severe anxiety.

SECONDARY OUTCOMES:
Thinc-it cognitive function test | basline、12weeks、24weeks
  The THINC-it tool is digitalized and completed by the respondent on a tablet is used to assess cognitive function in patients with MDD. Includes four objective test, Spotter (Choice Reactio Time), Symbol Check (1-back test), Trails (Trails Making Test B), and Codebreaker (Digit Symbol Substitution Test) as well as a self-reported cognitive function questionnaire (i.e., Perceived Deficit Questionnaire, 5-item).
Sheehan Disability Scale | basline、12weeks、24weeks
  It was used to evaluate the impairment of social function in three areas of work/school, social life and family life of patients with depression. 0～10 scores were used in each area, and the total score was 0～30 points. The higher the score, the more serious the impairment of function.
Pittsburgh Sleep Quality Index | baseline、2weeks、8weeks、12weeks、24weeks
  Using to assess the sleep quality. Total scores of 0-5 indicates that the quality of sleep is very good, 6～10 indicates that the quality of sleep is OK, 11～15 indicates that the quality of sleep is average, and 16～21 indicates that the quality of sleep is poor.
Gastrointestinal function scale | baseline、2weeks、8weeks、12weeks、24weeks
  A rating scale for gastrointestinal symptoms in patients. It contains 16 items, total scores 16～112, each items is graded on a scale of 1～7, the higher total scores, the more severe the gastrointestinal symptoms.

OTHER OUTCOMES:
Serum metabolites | baseline、2weeks、8weeks、12weeks、24weeks
  Metabolites in serum were quantified using LC-MS/MS. LC-MS/MS analyses were performed using a UHPLC system.
Shotgun Metagenomic Sequencing and Metagenome-Wide Intestinal macrogene | baseline、2weeks、8weeks、12weeks、24weeks
  Shotgun metagenomic sequencing and alignment methods were used to detect fecal flora diversity

CONTACTS AND LOCATIONS:
Overall Officials: Ma x c, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- 277 Yanta West Road, Xi'an, Yanta, China

IPD SHARING:
Plan to Share IPD: No